CLINICAL TRIAL: NCT03160482
Title: Evaluation of PACE4 Isoforms as Biomarkers in Thyroid Cancer
Brief Title: PACE4 in Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Robert Day (Other)
Responsible Party: Sponsor-Investigator, Robert Day, PhD, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Other Study IDs: 2017-1620
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Thyroid Nodule
Keywords: Thyroid Neoplasm; Thyroid Cancer; Bethesda Classification; Biomarkers; Protein convertase
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Formalin-fixed, paraffin-embedded thyroid tissue, kept at the CIUSSS de l'Estrie - CHUS Pathology archives
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Papillary carcinoma, classical variant
  Interventions: Diagnostic Test: Immunohistochemistry
- Follicular carcinoma
  Interventions: Diagnostic Test: Immunohistochemistry
- Colloid nodule
  Interventions: Diagnostic Test: Immunohistochemistry
- Hyperplastic nodule
  Interventions: Diagnostic Test: Immunohistochemistry
- Adenomatoid nodule
  Interventions: Diagnostic Test: Immunohistochemistry
- Follicular adenoma
  Interventions: Diagnostic Test: Immunohistochemistry
- Papillary carcinoma, follicular variant
  Interventions: Diagnostic Test: Immunohistochemistry
- Medullary carcinoma
  Interventions: Diagnostic Test: Immunohistochemistry
- Lymphocytic thyroiditis
  Interventions: Diagnostic Test: Immunohistochemistry

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry — Immunohistochemistry procedure on the formalin-fixed, paraffin-embedded tissue.

SUMMARY:
The investigation of thyroid nodules is limited by the fact that up to 49% of the fine needle aspirations (FNA) performed are of "indeterminate cytological signification". Moreover, no fully reliable molecular marker for thyroid cancer have been described. The goal of this project is to study the expression of a specific kind of protein convertase in benign and in malignant thyroid nodules to determine its potential as a biomarker.

DETAILED DESCRIPTION:
Patients that underwent thyroidectomy at the CIUSSS de l'Estrie-CHUS will be recruited and classified according to the pathological diagnosis. An immunohistochemistry technique, developed and calibrated for the specific protein convertase studied, will be undertaken. Results will be interpreted by a specialized pathologist.

ELIGIBILITY:
Inclusion Criteria:

* Men of women, aged 18-100 y.-o.
* History of subtotal or total thyroidectomy at the "Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre hospitalier universitaire de Sherbrooke" (CIUSSS de l'Estrie - CHUS) between January 2010 and May 2016.

Exclusion Criteria:

* Refusal to participate to the study.
* Unavailability of the formalin-fixed, paraffin-embedded tissues.
* Uncertain pathological diagnosis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the territory of the CIUSSS de l'Estrie - CHUS, that underwent a subtotal or total thyroidectomy
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Expression pattern of the studied protein convertase | Trough study completion, an average of 1 year after the patients have been operated.
  Horseradish peroxidase staining with specific antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Day, PhD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fradet L, Temmar R, Couture F, Belzile M, Fortier PH, Day R. Evaluation of PACE4 isoforms as biomarkers in thyroid cancer. J Otolaryngol Head Neck Surg. 2018 Oct 19;47(1):63. doi: 10.1186/s40463-018-0311-x. PMID 30340539